CLINICAL TRIAL: NCT03944668
Title: Comprehensive Cardiac Rehabilitation Feasibility After Stroke
Acronym: CCRFast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-361
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Results first posted 2021-02-24 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2020-09

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: single arm, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Exercise intervention
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 36 sessions of comprehensive cardiac rehabilitation over 12 weeks

SUMMARY:
Comprehensive Cardiovascular Rehabilitation Feasibility After Stroke (CCR FAST) will evaluate the feasibility of enrolling Regions Hospital stroke patients in a Comprehensive Cardiovascular Rehabilitation (CCR) program. CCR will include aerobic exercise and patient education (regarding risk factors and medication compliance), similar to the rehabilitation program for cardiac disease patients. The overall goal of CCR FAST is to demonstrate the feasibility and safety of including stroke patients in a CCR program, while examining the clinical value in reducing stroke recurrence, myocardial infarction, readmission, and mortality in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient has suffered an ischemic stroke
* Patient should be ambulatory (non-disabling stroke) to be able to participate in the CCR exercise program
* Patient is able to start cardiac rehabilitation within 2 weeks of stroke

Exclusion Criteria:

* No baseline (index admission for ischemic stroke) MRI completed
* Life expectancy < 1-year
* Presence of brain hemorrhage: intracerebral hemorrhage, subarachnoid hemorrhage, subdural hematoma, or epidural hematoma
* Concurrent diagnosis of seizure disorder
* Patient with moderate or severe neurologic deficits, limiting their ability to participate in the CCR exercise program
* Cardiopulmonary conditions preventing the patient from participation, such as severe heart failure, severe aortic stenosis, and exercise-induced asthma
* Patient with cognitive dysfunction impairing their ability to follow directions
* Anticipated procedures such as carotid stenting, carotid endarterectomy, and intracranial aneurysm coiling
* Patient unable to commit to the frequent visits of the CCR program
* Participation in other interventional research (observational research is allowed)
* Unable to have brain MRI
* Non-English speaker
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haitham M Hussein, MD, Principal Investigator — Regions Hospital Stroke Center
Locations (3):
- United States (3):
  - Regions Hospital, Saint Paul, Minnesota
  - Regions Hospital Outpatient Cardiopulmonary Rehabilitation Clinic, Saint Paul, Minnesota
  - HealthPartners Neuroscience Center, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 patients assessed for eligibility
  * 9 refused to participate
  * 6 unable to reach
Period: Overall Study
Arm/Group | Intervention
Started | 17 (Enrolled in Study)
Able to Use Patient Data | 14 (3 Patient's Data Unusable)
Participated in Intervention | 10 (Started Cardiac Rehabilitation)
Completed | 8 (Completed 75% of Comprehensive Cardiac Rehabilitation Sessions)
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: 14 Enrolled and consented stroke patients
Arm/Group | Intervention
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Smoking Status [Count of Participants; unit: Participants]
  Current | 4
  Previous | 3
  Never | 7
Stroke Mechanism [Count of Participants; unit: Participants]
  Cryptogenic | 3
  Cardiomebolic | 3
  Large Vessel Extracranial | 4
  Lacunar | 2
  Other/Missing | 2
National Institutes of Health Stroke Scale (NIHSS) [Median (Inter-Quartile Range); unit: units on a scale] — NIHSS is a tool used to evaluate stroke severity. The total score ranges from 0-42, with a higher score indicating a more severe stroke.
  units on a scale | 0.5 [0 to 1]
Length of Stay for Initial Stroke Admission [Mean (Standard Deviation); unit: days] | 1.8 (1.1)
Weight [Mean (Standard Deviation); unit: lbs] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  lbs
    number analyzed (Participants) | 10
    (all) | 220.2 (34.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  kg/m^2
    number analyzed (Participants) | 10
    (all) | 35.1 (8.0)
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mmHg
    number analyzed (Participants) | 10
    (all) | 136.9 (17.5)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mmHg
    number analyzed (Participants) | 10
    (all) | 78.9 (14.4)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program, had baseline physical visit, and got results from respective lab
  mg/dL
    number analyzed (Participants) | 9
    (all) | 188.4 (124.1)
HDL [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mg/dL
    number analyzed (Participants) | 10
    (all) | 39.6 (7.3)
LDL [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program, had baseline physical visit, and got results from respective lab
  mg/dL
    number analyzed (Participants) | 9
    (all) | 105.7 (36.2)
Non-HDL [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mg/dL
    number analyzed (Participants) | 10
    (all) | 139.1 (41.5)
Sodium [Mean (Standard Deviation); unit: mEq/L] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mEq/L
    number analyzed (Participants) | 10
    (all) | 138.1 (3.1)
Potassium [Mean (Standard Deviation); unit: mEq/L] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mEq/L
    number analyzed (Participants) | 10
    (all) | 4.0 (0.3)
Chloride [Mean (Standard Deviation); unit: mEq/L] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mEq/L
    number analyzed (Participants) | 10
    (all) | 103.9 (2.2)
Bicarbonate (cO2) [Mean (Standard Deviation); unit: mEq/L] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mEq/L
    number analyzed (Participants) | 10
    (all) | 24.1 (3.5)
Glucose [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mg/dL
    number analyzed (Participants) | 10
    (all) | 141.9 (82)
Creatinine [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mg/dL
    number analyzed (Participants) | 10
    (all) | 1.0 (0.2)
Calcium [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mg/dL
    number analyzed (Participants) | 10
    (all) | 9.4 (0.6)
Anion Gap [Mean (Standard Deviation); unit: mEq/L] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  mEq/L
    number analyzed (Participants) | 10
    (all) | 10.4 (1.7)
International Normalized Rate (INR) [Mean (Standard Deviation); unit: ratio] — Population: Only patients who began CCR Fast exercise program, had baseline physical visit, and got results from respective lab
  ratio
    number analyzed (Participants) | 7
    (all) | 1.0 (0.1)
Prothrombin Time (PT) [Mean (Standard Deviation); unit: seconds] — Population: Only patients who began CCR Fast exercise program, had baseline physical visit, and got results from respective lab
  seconds
    number analyzed (Participants) | 6
    (all) | 25.9 (6.6)
A1c [Mean (Standard Deviation); unit: mg/dL] — Population: Only patients who began CCR Fast exercise program, had baseline physical visit, and got results from respective lab
  mg/dL
    number analyzed (Participants) | 8
    (all) | 7.8 (3.6)
Glomerular Filtration Rate [Count of Participants; unit: Participants] — Population: Only patients who began CCR Fast exercise program and had baseline physical visit
  Participants
    number analyzed (Participants) | 10
    > 60 | 7
    < 60 | 3

OUTCOME MEASURES:

1. Primary Outcome: Attendance Rate
Description: 75% attendance at comprehensive cardiovascular rehabilitation (CCR) sessions
Time Frame: 12 weeks
Population: 14 Stroke patients who enrolled and consented in study
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants | 8

2. Secondary Outcome: Number of Patients With or Without Recurrent Stroke
Description: Recurrent stroke in follow-up period
Time Frame: 6 month
Population: 14 Stroke patients who enrolled and consented in study
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Stroke patients enrolled in study
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants
  No recurrent stroke | 8
  Lost to follow-up | 6

3. Secondary Outcome: Number of Participants With or Without Myocardial Infarction
Description: Myocardial infarction in follow-up time
Time Frame: 6 month
Population: 14 Stroke patients who enrolled and consented in study
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants
  No myocardial infarction | 8
  Lost to follow-up | 6

4. Secondary Outcome: Hospital Readmission
Description: rate, for a cardiovascular or cerebrovascular indication
Time Frame: 6 month
Population: 14 Stroke patients who enrolled and consented in study
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants
  No | 8
  Lost to follow-up | 6

5. Secondary Outcome: Number of Participants With or Without Silent Stroke
Description: rate, on MRI
Time Frame: 6 month
Population: 14 Stroke patients who enrolled and consented in study
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants
  Yes, silent stroke | 1
  No silent stroke | 7
  Lost to follow-up | 6

6. Secondary Outcome: Number of Participants Without Death
Description: rate
Time Frame: 6 month
Population: 14 Stroke patients who enrolled and consented in study
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 14
Participants
  No death | 8
  Lost to follow-up | 6

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/68/NCT03944668/Prot_SAP_000.pdf